CLINICAL TRIAL: NCT00255385
Title: Evaluating Efficacy of Milk Fortified With Bifidus DR10-Oligosaccharides, Zinc and Iron in Reducing Morbidity Due to Diarrhea, Pneumonia and Improving Growth and Development in Children Ages 13-36 Months
Brief Title: Efficacy of Bifidus DR10 and Oligo Saccharides / Micronutrient Fortification of Milk
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Annamalai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H22010703A
Record Dates: First submitted 2005-11-16; First posted 2005-11-18 (Estimated); Last update posted 2005-11-18 (Estimated); Status verified 2005-04

CONDITIONS: Diarrhea; Pneumonia; Febrile Illness; Growth; Child Development
Keywords: Zinc; Iron; Probiotics; Prebiotics; Child health; Milk fortification; Randomized controlled trial
MeSH Terms: conditions — Diarrhea; Pneumonia | interventions — Micronutrients; Zinc; Iron; Lead

INTERVENTIONS:
Drug: Micronutrient (Zinc and Iron) fortification
Drug: Pre and Probiotic fortification

SUMMARY:
The purpose of the study is to evaluate effect or fortifying milk with pre and probiotics or with micronutrients on prevention of diarrhea, pneumonia and other childhood illnesses and improvement in growth and development.

DETAILED DESCRIPTION:
The 1993 World Bank World Development Report (1) delivered a strong but sad reminder of the dramatic scale of suffering and death among preschool children attributable to pneumonia (2.7million in 1990) and diarrhea (another 2.5million deaths). In terms of "disability adjusted life years" (DALYS) lost, in 0-4 years old children, respiratory infections account for 18.5% and 17.6% (in boys & girls respectively) and diarrhea accounts of another 16.2% and 15.7% respectively. The development of effective interventions to reduce morbidity from these illnesses has become a humanitarian, economic and political imperative and essential in achieving the morbidity and mortality reduction goals that the "World Summit for Children" set a decade ago. Therapy with Oral Rehydration Solution (ORS) for diarrhea, a cornerstone of the universal strategy for child survival, has low compliance due to having no effect on duration of diarrhea and has mixed impact on child mortality (2-5). Present strategies for containing morbidity and mortality due to respiratory infection focuses primarily on antibiotic treatment. Increasing prevalence of antibiotic resistant strains, poses a problem with the current strategy. Lack of any truly effective and affordable preventive vaccine, for both diarrhea and pneumonia has aroused considerable interest in food based preventive interventions. In the recent years increasing recognition and evidence regarding the role of Probiotics, and micronutrients like Zinc, as both preventive and therapeutic agents against infections has made them a potential and promising candidate. This study is in fact two trial run concurrently with two milk preparation one fortified with pre and Probiotics and second fortified with micronutrients and each having same milk unfortified as control.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12-36 months at enrollment
* Resident of Sangam Vihar and likely to be in the area for 1 year.
* Parents consenting to participate in the trial.

Exclusion Criteria:

* Children who have been given complete therapeutic/preventive course of Iron in the last 6 months.
* Children currently as part of a different Iron/Zinc supplementation program.
* Children known to be allergic to milk.
* Children who are severely malnourished and requiring hospitalization.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200
Dates: Start 2002-04; Study Completion 2004-04

PRIMARY OUTCOMES:
Diarrhea
Pneumonia
Febrile illness
Growth
Development
Activity

SECONDARY OUTCOMES:
Iron status
Zinc status
Colonization
Copper status

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sazawal, MD, MPH, PHD, Principal Investigator — Johns Hopkins University; VenuGopal P Menon, PhD, Principal Investigator — Annamalai University; Robert E Black, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Center for Micronutrient Research, New Delhi, New Delhi, India

REFERENCES:
- [Derived] Sazawal S, Dhingra U, Dhingra P, Dutta A, Shabir H, Menon VP, Black RE. Efficiency of red cell distribution width in identification of children aged 1-3 years with iron deficiency anemia against traditional hematological markers. BMC Pediatr. 2014 Jan 15;14:8. doi: 10.1186/1471-2431-14-8. PMID 24428927
- [Derived] Sazawal S, Dhingra U, Dhingra P, Hiremath G, Sarkar A, Dutta A, Menon VP, Black RE. Micronutrient fortified milk improves iron status, anemia and growth among children 1-4 years: a double masked, randomized, controlled trial. PLoS One. 2010 Aug 13;5(8):e12167. doi: 10.1371/journal.pone.0012167. PMID 20730057
- [Derived] Sazawal S, Dhingra U, Hiremath G, Sarkar A, Dhingra P, Dutta A, Verma P, Menon VP, Black RE. Prebiotic and probiotic fortified milk in prevention of morbidities among children: community-based, randomized, double-blind, controlled trial. PLoS One. 2010 Aug 13;5(8):e12164. doi: 10.1371/journal.pone.0012164. PMID 20730056
- [Derived] Sazawal S, Dhingra U, Dhingra P, Hiremath G, Kumar J, Sarkar A, Menon VP, Black RE. Effects of fortified milk on morbidity in young children in north India: community based, randomised, double masked placebo controlled trial. BMJ. 2007 Jan 20;334(7585):140. doi: 10.1136/bmj.39035.482396.55. Epub 2006 Nov 28. PMID 17132678